CLINICAL TRIAL: NCT04580251
Title: Ideal Marker for Targeted Axillary Dissection
Acronym: IMTAD
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Collaborators: Silesian Hospital in Opava (Other); Masaryk Memorial Cancer Institute (Other); EUC Clinic in Zlín (Unknown); Institute for the Care of Mother and Child, Prague, Czech Republic (Other); University of Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: CHIR-05-IMTAD
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer
Keywords: breast cancer; axillary dissection; Magseed marker; iodine seed; carbon suspension; axillary lymph node
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Magnetic marker Magseed: Patients in whom the magnetic marker Magseed is used will be enrolled in this study arm and will undergo targeted axillary dissection.
  Interventions: Procedure: Targeted axillary dissection
- Iodine seed 125I marker: Patients in whom the iodine seed 125I marker is used will be enrolled in this study arm and will undergo targeted axillary dissection.
  Interventions: Procedure: Targeted axillary dissection
- Carbon suspension: Patients in whom the carbon suspension marker is used will be enrolled in this study arm and will undergo targeted axillary dissection.
  Interventions: Procedure: Targeted axillary dissection

INTERVENTIONS:
Procedure: Targeted axillary dissection — The surgical treatment procedure of targeted axillary dissection performed in patients in whom the pathological lymph nodes have been marked using the examined and compared markers (magnetic marker Magseed, iodine seed 125I, carbon suspension)

SUMMARY:
A multicentre prospective comparative study, comparing the use of various markers (magnetic marker Magseed, iodine seed 125I, carbon suspension) for marking a pathological lymph node in patients with breast carcinoma prior to neoadjuvant therapy and subsequent surgical treatment consisting of targeted axillary dissection.

DETAILED DESCRIPTION:
There are two basic aims of the study

1. Prospective comparison of the reliability and accuracy of individual markers used for marking of a pathological axillary lymph node with subsequent targeted axillary dissection.
2. Comparison of the number of complications during localizing and detection of individual markers and postoperative complications.

In individual collaborating centers, these markers are commonly used in clinical practice for marking of a pathological lymph node in patients with breast carcinoma. The usual standard of practice and treatment will not be changed in any way; the patients will only be prospectively followed. The study will bring an answer to the question of which marker is the best for marking lymph nodes.

Apart from the basic demographic and other data (patient age, side of the body, size and characteristics of the tumor (typing, grading, staging), type and time of surgery, the incidence of complications during implantation or detection of the marker, number of lymph nodes, complications after surgery, and the final histological findings, also the following outcome measures will be observed:

* depth of marker implantation (measured in mm)
* marker migration (measured in mm)
* success-rate of resection of the marked lymph node - assessment, whether the lymph node was removed (yes/no) using the respective marker, expressed in percent of successful removal for the respective marker
* time from localizing the pathological lymph node using the marker to surgery (measured n days)

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of breast cancer, confirmed with a biopsy
* indication of neoadjuvant therapy
* biopsy of pathologically enlarged axillary lymph node and marking of the lymph node using one of the markers before neoadjuvant chemotherapy
* surgical treatment after neoadjuvant chemotherapy (targeted axillary dissection)

Exclusion Criteria:

* refusal to participate in the study
* another treatment protocol, which does not include targeted axillary dissection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with breast cancer confirmed with a biopsy, indicated for neoadjuvant chemotherapy and axillary dissection, in whom pathological lymph nodes have been marked using one of the three examined and compared markers.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Depth of marker implantation | During surgery/intervention
  The depth of marker implantation will be assessed and measured in millimetres
Marker migration | During surgery/intervention
  Marker migration will be assessed and measured in millimetres
Success-rate of resection of the marked lymph node | 1 month
  Assessment, whether the lymph node was removed (yes/no) using the respective marker, expressed in percent of successful removal for the respective marker.
Time from localizing the pathological lymph node using the marker to surgery | 1 month
  The time from localizing the pathological lymph node using the marker to surgery will be analysed and measured in days

CONTACTS AND LOCATIONS:
Overall Officials: Jan Žatecký, MD, Principal Investigator — Silesian Hospital in Opava
Locations (5):
- Czechia (5):
  - Silesian Hospital in Opava, Opava, Moravian-Silesian Region
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region
  - Institute for the Care of Mother and Child, Prague, Czech Republic, Prague, Prague
  - Masaryk Memorial Cancer Institute, Brno, South Moravian
  - EUC Clinic in Zlín, Zlín, Zlín

IPD SHARING:
Plan to Share IPD: No
Individual participant data may be made available to other researchers upon request.

REFERENCES:
- [Derived] Zatecky J, Coufal O, Zapletal O, Kubala O, Kepicova M, Faridova A, Raus K, Gatek J, Kosac P, Peteja M. Ideal marker for targeted axillary dissection (IMTAD): a prospective multicentre trial. World J Surg Oncol. 2023 Aug 19;21(1):252. doi: 10.1186/s12957-023-03147-x. PMID 37596658